CLINICAL TRIAL: NCT04430868
Title: The Impact of Lifestyle Redesign Program in Schizophrenia
Brief Title: Lifestyle Redesign For Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taoyuan Psychiatric Center, Ministry of Health and Welfare, Executive Yuan, R.O.C. Taiwan (Other Government)
Responsible Party: Principal Investigator, YU SHIUAN LIAW, Occupational Therapist, Taoyuan Psychiatric Center, Ministry of Health and Welfare, Executive Yuan, R.O.C. Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B20190705
Record Dates: First submitted 2020-06-11; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Schizophrenia; Rehabilitation
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LRP group (Experimental): The participants in LRP group receive lifestyle redesign program plus treatment as usual. The LRP intervention consisted of one 90-minute session each week for 10 weeks
  Interventions: Behavioral: lifestyle redesign program
- TAU group (No Intervention): The participants in TAU group received usual treatment at the same time as LRP group.

INTERVENTIONS:
Behavioral: lifestyle redesign program — In this group, it starts with health education, the participants then change their opinions and experience health activities, and it ends with discussion and sharing their experience.
  Arms: LRP group

SUMMARY:
This study aimed to investigate the effects of lifestyle redesign program plus treatment as usual versus treatment as usual on cognition, psychiatric symptoms, quality of life, and occupational engagement for schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia, based on the ICD-10 diagnostic criteria for research (World Health Organization, 1992)
* age from 20 to 65
* attending day care center regularly for at least 1 month and taking stable dose of medication

Exclusion Criteria:

* comorbid other mental disorder (e.g. depression, anxiety, ADHD...etc.)
* comorbid mental retardation
* lacking the reading and writing skills

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Change scores of Brief Psychiatric Symptom Rating Scale (BSRS) | 3 times: 1 to 2 weeks before intervention, 1 to 5 days after intervention and at 1 month after intervention
  The Chinese version of BSRS with 50 items is administered to measure psychiatric symptoms. BSRS items were evaluated on a five-point Likert scale from 0 (not present) to 4 (extremely severe). The total score ranged from 0 to 200, with higher scores reflecting more severe of psychiatric symptoms.
Change scores of Occupational Self Assessment (OSA) | 3 times: 1 to 2 weeks before intervention, 1 to 5 days after intervention and at 1 month after intervention
  The OSA with 29 items is administered to measure occupational engagement.
Change scores of Schizophrenia Quality of Life Scale Revision 4 (SQLS-R4) | 3 times: 1 to 2 weeks before intervention, 1 to 5 days after intervention and at 1 month after intervention
  The Chinese version of Schizophrenia Quality of Life Scale Revision 4 (SQLS-R4) was administered to measure subjective quality of life. The total scores ranged from 33-165, with higher scores indicating comparatively lower quality of life.
Change scores of Montreal Cognitive Assessment (MoCA) | 3 times: 1 to 2 weeks before intervention, 1 to 5 days after intervention and at 1 month after intervention
  The Chinese version of MoCA was administered to measure cognition, with higher scores indicating better cognition.